CLINICAL TRIAL: NCT00235625
Title: A Phase II Open Label Study of the Safety and Efficacy of Curcuminoids C3 Complex® in Patients With Chronic Psoriasis Vulgaris.
Brief Title: Curcuminoids for the Treatment of Chronic Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 803489
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Psoriasis
Keywords: Alternative Medicine; Psoriasis; Turmeric; Curcumin; Dermatology
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Curcuminoids C3 Complex®

SUMMARY:
Turmeric (Curcuma Longa) is member of the ginger family and is best known for its culinary use as the major of component of curry powder. The volatile of oils (called curcuminoids) of the turmeric root, however, have anti-inflammatory actions which make them promising candidates for the treatment of psoriasis. For example, curcumin has been shown to improve psoriasis in experiments using in vitro models. Turmeric has been shown to have minimal side effects in doses up to 12 grams per day. The purpose of this study is to determine the safety and to estimate the efficacy of oral Curcuminoid C3 Complex® in patients with chronic psoriasis vulgaris.

DETAILED DESCRIPTION:
This study is no longer recruiting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have chronic plaque type psoriasis that, in the investigator's opinion is clinically stable and does not require urgent treatment with standard, FDA approved psoriasis therapies.
* Psoriasis must cover at least 6% of subject's body surface area and lesions must have moderate plaque thickness
* Subjects must be willing to and have the capacity for giving written informed consent
* Ages 18 to 75
* Subjects must be available for the total duration of the study (16 weeks)
* Female subjects that are sexually active with male partners must be postmenopausal, surgically incapable of childbearing, or be using a medically acceptable method of contraception throughout the entire study period. Medically acceptable methods of contraception that may be used by the subject and/or partner include oral contraceptives or patch, diaphragms with spermicide, IUD, condom with spermicide, or progestin implant or injection. Females taking oral contraceptives must have taken them consistently for at least two months prior to receiving study medication. All female subjects must consent to a urine pregnancy test at screening and at start of study, which must be negative at both time points. Male subjects who are sexually active with female partners and are capable of fertilization must ensure that their female partners will either be postmenopausal, surgically incapable of childbearing, or will use a medically acceptable method of contraception throughout the entire study period

Exclusion Criteria:

•Females subjects who are pregnant or nursing a child •Subjects who are sensitive to or allergic to turmeric or curry powder •History of alcohol or drug abuse within 12 months of screening visit •Subjects with rapidly improving or deteriorating psoriasis or the following more variable types of psoriasis: guttate, erythrodermic, or pustular psoriasis •Use of systemic treatments for psoriasis (including methotrexate, cyclosporine, alefacept, adalimumab, efalizumab, infliximab, etanercept, etretinate, systemic steroids and PUVA) within 3 months prior to day 0 or at any time during the study. •Use of topical treatments and UVB therapy for psoriasis (not including non-medicated emollients or shampoos) within 14 days prior to day 0 or at any time during the study period. •Subjects, who have received an experimental drug, used any experimental medical devise within 30 days prior to screening •Clinically significant laboratory abnormalities •Subjects with significant medical comorbidities •Subjects for whom the dose of the following medications has changed within 1 month of day 0: clonidine, digoxin, beta-blockers, lithium, or anti-malarials •Subjects unable to swallow pills •Subject who are unable to adhere to the protocol for any reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-10; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Physicians Global Assessment (PGA) of Change | November 2007

SECONDARY OUTCOMES:
PASI (Psoriasis Area Severity Index) | November 2007
quality of life (Skindex-29) | November 2007
pharmacodynamic activity (via skin biopsies and serum cytokines) | December 2007

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Gelfand, MD/MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States